CLINICAL TRIAL: NCT01741272
Title: Early Mobilization Following Mini-Open Rotator Cuff Repair: A Randomized Clinical Trial
Brief Title: Early Mobilization Following Mini-Open Rotator Cuff Repair
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00001096
Record Dates: First submitted 2012-11-29; First posted 2012-12-04 (Estimated); Results first posted 2015-03-17 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Full Thickness Rotator Cuff Tears
Keywords: rotator cuff tear; arthroscopically assisted; health related quality of life(HRQL); functional outcome
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Suburethral Slings

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Usual Care) (Active Comparator): Will be immobilized in a sling for 6 weeks. Intervention: Procedure: Sling
  Interventions: Procedure: Sling
- Group B (Early ROM) (Experimental): Will use the sling for comfort only. Intervention: Procedure: No sling
  Interventions: Procedure: No sling

INTERVENTIONS:
Procedure: Sling — Patients will use a sling for 6 weeks as per usual care. No active ROM allowed.
  Arms: Group A (Usual Care)
Procedure: No sling — Patients may discontinue use of the sling as early as pain and comfort allow. Early active ROM is allowed for activities of daily living.
  Arms: Group B (Early ROM)

SUMMARY:
The primary objective of this study is to determine if early active range of motion after mini-open rotator cuff repair in adults results in improved shoulder range of motion at 6 weeks and 3 months after surgery. The secondary objective of this study is to determine if early mobilization improves disease-specific quality of life and promotes earlier return to work/function.

Hypothesis: Adults undergoing mini-open rotator cuff repair will have faster recovery of range of motion, improved disease specific quality of life and earlier return to work/function if allowed to begin early active range of motion compared to subjects who are immobilized in a sling for 6 weeks.

DETAILED DESCRIPTION:
The rotator cuff is a group of four muscles around the shoulder. They function to provide both shoulder mobility and power as well as stability. Rotator cuff tears can be a significant cause of pain and disability for the patient. Surgical repair is done to reconnect the torn tendon(s) to the bone and has been shown to be an effective treatment in the presence of full-thickness tears. The goals of Rotator Cuff (RC)surgery are to decrease pain, increase range of motion(ROM) and strength. This is done with a small incision called a mini-open. Standard care following this surgical repair is to be placed in a sling for 6 weeks to protect the repaired shoulder tendons. During this time ROM exercises are done using the non-operated arm for assistance. No active or voluntary movement is allowed during the first 6 weeks. Unfortunately, some of these patients develop shoulder stiffness which slows their recovery and return to work or daily activities and may result in increased use and cost of rehabilitation services.

The purpose of this study is to determine if following a RC repair, patients can safely stop wearing their sling and begin active ROM for activities of daily living as early as pain and comfort allow. A total of 190 patients have been recruited to this study (95/group) were randomly assigned to one of two study groups. Patients in Group A (sling for 6 weeks) will wear their sling for 6 weeks. Self-assisted ROM exercises are allowed at any time, but active movement will not be allowed until 6 weeks after surgery. Patients in Group B (Sling as needed) will be allowed to remove their sling as early as pain and comfort allow. Self-assisted ROM exercises are allowed at any time as are active ROM for activities of daily living. Patients who agree to participate will be seen by their surgeon and the research coordinator for a baseline assessment before surgery and again at 2 & 6 weeks, 3, 6, 12 and 24 months after surgery. Each visit will include a ROM assessment and disease specific quality of life questionnaires. Patients will also undergo an Ultrasound exam at a minimum of 2 years after surgery to verify the integrity of their RC repair. Differences in ROM, questionnaire scores, RC integrity and adverse events will be examined between the two groups.

ELIGIBILITY:
Inclusion Criteria:

Clinical:

* males and females over 18 years of age
* failed non-operative management defined as persistent pain and/or disability following 3 months of conservative medical treatment including analgesic/anti-inflammatory medications, intra-articular corticosteroids, activity modification and physical therapy.

Radiological:

* confirmed full-thickness rotator cuff tear on arthrogram or MRI

Surgical:

* full-thickness tear of the rotator cuff confirmed through arthroscopy
* rotator cuff repairable using mini-open approach

Exclusion Criteria:

* previous shoulder surgery
* previous fracture of scapula or humerus
* history of charcot joint or inflammatory arthropathy
* cervical radiculopathy
* active joint or systemic infection
* neurological disorder
* significant paralysis of the rotator cuff, deltoid or shoulder girdle musculature
* major medical illness (life expectancy less than 2 years or unacceptably high operative risk)
* unable to speak or read English
* immunosuppressive therapy or chronic steroids (eg. prednisone)
* patient unwilling to be followed for 2 years
* psychiatric illness that precludes informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2003-09; Primary Completion 2013-01 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Balyk, MD, FRCSC, Principal Investigator — University of Alberta
Locations (1):
- Grey Nuns Community Hospital, Edmonton, Alberta, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A (Usual Care) | Group B (Early ROM)
Started | 92 | 97
Completed | 92 | 97
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No significant differences in baseline characteristics. Mean age: Group A 54.9(35;78), Group B 55.4(38;86). Males (%): Group A 58(63), Group B 57(58.8).
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A (Usual Care) | Group B (Early ROM) | Total
Number analyzed (Participants) | 92 | 97 | 189
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 54.9 [35 to 78] | 55.4 [38 to 86] | 55.1 [35 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 40 | 74
  Male | 58 | 57 | 115
Region of Enrollment [Number; unit: participants]
  Canada | 92 | 97 | 189

OUTCOME MEASURES:

1. Primary Outcome: Change in Range of Motion (ROM)From Baseline to 24 Months
Description: Two-way repeated-measures analysis of variance (ANOVA) compared shoulder ROM between groups over time. Standing: Active flexion, scaption, abduction, extension, internal rotation (vertebral level).
  Supine Lying: Active and passive flexion, abduction, external rotation (arm at side), external rotation (arm at 90 degrees abduction), internal rotation (arm at side), internal rotation (arm at 90 degrees abduction),and horizontal adduction.
Time Frame: Baseline, 6 weeks, 3, 6, 12, 24 months
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Group A (Usual Care) | Group B (Early ROM)
Number analyzed (Participants) | 92 | 97
degrees
  Baseline Forward Flexion | 124.4 (33.9) | 120.2 (30.2)
  6 weeks Forward Flexion | 73.2 (32.1) | 84.1 (30.2)
  3 months Forward Flexion | 118.5 (25.5) | 120.0 (25.4)
  6 months Forward Flexion | 135.9 (21.6) | 136.3 (18.1)
  12 months Forward Flexion | 144.8 (19.2) | 144.8 (12.4)
  24 months Forward Flexion | 149.6 (17.8) | 149.9 (12.4)
  Baseline Abduction | 117.4 (40.1) | 116.3 (40.3)
  6 weeks Abduction | 68.5 (27.8) | 81.4 (26.3)
  3 months Abduction | 113.0 (26.2) | 112.1 (29.1)
  6 months Abduction | 139.1 (25.8) | 134.6 (27.3)
  12 months Abduction | 149.9 (23.2) | 144.7 (22.6)
  24 months Abduction | 155.5 (20.2) | 150.7 (20.0)
  Baseline External Rotation in Abduction | 65.2 (35.6) | 56.9 (36.2)
  6 weeks External Rotation in Abduction | 15.0 (28.2) | 22.6 (29.1)
  3 months External Rotation in Abduction | 53.7 (26.9) | 52.6 (29.1)
  6 months External Rotation in Abduction | 74.2 (17.1) | 73.1 (17.3)
  12 months External Rotation in Abduction | 80.3 (13.9) | 77.9 (13.4)
  24 monthsExternal Rotation in Abduction | 84.0 (11.9) | 81.5 (11.7)
  Baseline Internal Rotation in Abduction | 30.7 (19.9) | 26.7 (19.2)
  6 weeks Internal Rotation in Abduction | 7.7 (14.4) | 11.9 (16.1)
  3 months Internal Rotation in Abduction | 24.1 (13.8) | 23.7 (16.0)
  6 months Internal Rotation in Abduction | 32.9 (12.0) | 32.2 (12.7)
  12 months Internal Rotation in Abduction | 34.8 (10.3) | 33.9 (9.9)
  24 months Internal Rotation in Abduction | 35.7 (10.2) | 34.9 (9.7)
  Baseline Horizontal Adduction | 16.9 (14.2) | 14.4 (11.1)
  6 weeks Horizontal Adduction | 5.9 (9.1) | 6.4 (7.5)
  3 months Horizontal Adduction | 14.2 (9.7) | 12.5 (10.4)
  6 months Horizontal Adduction | 17.6 (9.0) | 16.2 (8.4)
  12 months Horizontal Adduction | 17.1 (8.0) | 17.5 (7.9)
  24 months Horizontal Adduction | 15.1 (6.0) | 15.2 (6.9)
  Baseline Scaption | 123.8 (36.1) | 125.1 (31.5)
  6 weeks Scaption | 72.1 (31.8) | 86.1 (30.7)
  3 months Scaption | 121.6 (26.9) | 122.2 (24.4)
  6 months Scaption | 140.3 (22.1) | 139.6 (20.2)
  12 months Scaption | 149.1 (18.4) | 146.6 (17.0)
  24 months Scaption | 151.0 (17.7) | 150.4 (13.3)

2. Secondary Outcome: Pain Questionnaire
Description: Shoulder pain was assessed using a visual analogue scale (VAS) where zero equals no pain and 10 is the worst possible pain at rest and with activity. Two-way repeated-measures analysis of variance (ANOVA) compared pain between groups over time.
Time Frame: Baseline, 2 weeks, 6 weeks, 3, 6, 12, 24 months
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Group A (Usual Care) | Group B (Early ROM)
Number analyzed (Participants) | 92 | 97
centimeters
  Baseline Pain at rest | 4.0 (2.8) | 4.0 (2.8)
  6 weeks Pain at rest | 2.3 (2.0) | 2.4 (2.5)
  3 months Pain at rest | 1.3 (1.6) | 1.4 (1.6)
  6 months Pain at rest | 0.93 (1.6) | 0.78 (1.3)
  12 months Pain at rest | 0.85 (1.7) | 0.49 (0.81)
  24 months Pain at rest | 0.53 (1.3) | 0.41 (0.89)
  Baseline Pain with activity | 5.2 (2.8) | 5.5 (3.1)
  6 weeks Pain with activity | 4.0 (2.3) | 3.3 (2.1)
  3 months Pain with activity | 2.8 (2.4) | 2.4 (2.0)
  6 months Pain with activity | 1.8 (2.2) | 1.6 (2.0)
  12 months Pain with activity | 1.1 (1.9) | 1.1 (1.4)
  24 months Pain with activity | 0.74 (1.4) | 0.81 (1.4)

3. Secondary Outcome: WORC Questionnaire
Description: Health related quality of life was measured using the Western Ontario Rotator Cuff Index (WORC). It is a 21-item disease specific questionnaire representing five quality of life domains (physical symptoms, sports and recreation, work, lifestyle and emotions). Each response is marked on a 100mm line in a VAS format with a maximum raw score of 2100, where zero represents the best and 2100 the worst score. This score is transformed to a 0-100 format, with 100 representing full shoulder function.
Time Frame: Baseline, 6, 12, 24 months
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | Group A (Usual Care) | Group B (Early ROM)
Number analyzed (Participants) | 92 | 97
units on a scale
  Baseline WORC Score | 40.1 [4.5 to 87] | 40.1 [2.4 to 86.6]
  24 months WORC Score | 90.9 [15.7 to 100] | 89.4 [48.4 to 100]

4. Secondary Outcome: Abduction Strength Using the Power Component of the Constant Score
Description: The Constant Score is the most widely used shoulder evaluation questionnaire in Europe and is a shoulder specific instrument. The score is a combination of an objective physical examination (65 points) and a subjective patient self evaluation (35 points). The physical examination component includes a range of motion assessment (forward elevation, lateral elevation, internal rotation, and external rotation) worth a total of 40 points (maximum of 10 points for each motion). The remaining 25 points are attributed to the strength assessment, where patients are awarded one point for each pound of pull that the patient can resist in abduction. Therefore the total possible score on the Constant score is 100 points (best possible score = 100. In this case only the power component was used therefore the best score is 25.
Time Frame: Baseline, 24 months
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | Group A (Usual Care) | Group B (Early ROM)
Number analyzed (Participants) | 92 | 97
units on a scale
  Mean Constant Power - Baseline | 8.7 [0 to 25] | 8.3 [0 to 25]
  Mean Constant Power - 24 months | 16.5 [0 to 25] | 16.3 [0 to 25]

5. Secondary Outcome: Complications
Description: Incidence of any surgical or medical complications will be prospectively documented.
Time Frame: 2 & 6 weeks, 3, 6, 12, 24 months
Population: 37 subjects (17 Early Mobilization, 20 Standard Rehabilitation) had non-re-tear complications. 5 subjects reported more than one complication.
Measure: Number; unit: participants
Arm/Group | Group A (Usual Care) | Group B (Early ROM)
Number analyzed (Participants) | 92 | 97
participants | 20 | 17

ADVERSE EVENTS:
Arm/Group | Group A (Usual Care) | Group B (Early ROM)
Serious Adverse Events (participants affected / at risk) | 0/92 | 0/97
Other Adverse Events (participants affected / at risk) | 20/92 | 17/97
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (Usual Care) (N=92) | Group B (Early ROM) (N=97)
Non re-tear complications (Musculoskeletal and connective tissue disorders) | 20 | 17 — all complications (pain, stiffnes, infection etc) were listed as a non re-tear complication and were not divided into seperate categories.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No